CLINICAL TRIAL: NCT00795002
Title: Randomized Phase II Study Comparing Two Administration Schedules of Flavopiridol (Alvocidib, NSC 649890, IND 46, 211) Given in Timed Sequential Combination With Cytosine Arabinoside (Ara-C) and Mitoxantrone Hydrochloride for Adults With Newly Diagnosed, Previously Untreated, Poor Risk Acute Myelogenous Leukemias (AML)
Brief Title: Alvocidib, Cytarabine, and Mitoxantrone in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00298; NCI-2009-00298 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000625222; J0856 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 8237 (Other: CTEP); P30CA006973 (NIH); U01CA070095 (NIH)
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — alvocidib; Mitoxantrone; Cytarabine

ARMS (2):
- Arm I (Experimental): Patients receive alvocidib IV over 1 hour on days 1-3, cytarabine IV continuously over 72 hours on days 6-8, and mitoxantrone hydrochloride IV over 60-120 minutes on day 9.
  Interventions: Drug: alvocidib; Drug: mitoxantrone hydrochloride; Drug: cytarabine; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm II (Experimental): Patients receive alvocidib IV over 30 minutes followed by alvocidib IV over 4 hours on days 1-3. Patients also receive cytarabine and mitoxantrone hydrochloride as in arm I.
  Interventions: Drug: alvocidib; Drug: mitoxantrone hydrochloride; Drug: cytarabine; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Novantrone
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying two different schedules of alvocidib to compare how well they work when given together with cytarabine and mitoxantrone in treating patients with newly diagnosed acute myeloid leukemia. Drugs used in chemotherapy, such as alvocidib, cytarabine, and mitoxantrone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not yet known which schedule of alvocidib is more effective when given together with cytarabine and mitoxantrone in treating patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the efficacy of two different schedules (bolus vs "hybrid bolus-infusion") of alvocidib followed by cytarabine and mitoxantrone hydrochloride in patients with newly diagnosed acute myeloid leukemia (AML) with poor-risk features.

SECONDARY OBJECTIVES:

I. To compare the toxicities of these regimens. II. To determine the disease-free survival and overall survival of patients who demonstrate a response to these regimens.

III. To compare the pharmacokinetics of alvocidib when administered in two different schedules (bolus vs "hybrid bolus-infusion").

IV. To describe alvocidib-induced alterations in AML blast cell expression of selected target mRNA and proteins.

V. To describe alvocidib-induced alterations in AML blast cell growth kinetic parameters.

OUTLINE: This is a multicenter study. Patients are stratified according to antecedent hematologic disorder of >= 6 months duration prior to transformation to acute myeloid leukemia (AML) and any prior antecedent therapy for myelodysplastic syndromes or myeloproliferative disorder. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive alvocidib IV over 1 hour on days 1-3, cytarabine IV continuously over 72 hours on days 6-8, and mitoxantrone hydrochloride IV over 60-120 minutes on day 9.

ARM II: Patients receive alvocidib IV over 30 minutes followed by alvocidib IV over 4 hours on days 1-3. Patients also receive cytarabine and mitoxantrone hydrochloride as in arm I.

Patients achieving partial or complete response (CR) after the first course of treatment may receive a second course of treatment 35-63 days following blood count recovery and/or undergo allogeneic bone marrow transplantation. Patients >= 50 years of age with t (8;21), inv (16), or t(16;16) AML who achieve CR after the first course of treatment may receive 3-4 courses of high-dose cytarabine consolidation therapy.

Bone marrow and/or blood samples are collected at baseline and periodically during study for correlative laboratory studies, including pharmacokinetic studies by liquid chromatography and tandem mass spectrometry, analysis of blast cell growth kinetic parameters by flow cytometry, and blast cell expression of selected target mRNA and protein by quantitative RT-PCR and western blotting.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed newly diagnosed acute myeloid leukemia (AML) meeting the following criteria:

  * Subtypes M0, M1, M2, M4-7
  * No acute promyelocytic leukemia (M3)
* At least 50 years of age OR >= 18 years of age with >= 1 of the following poor-risk disease features:

  * Antecedent hematologic disorder, including myelodysplastic syndromes (MDS)-related AML or prior myeloproliferative disorder (MPD)
  * Treatment-related AML, AML with trilineage dysplasia
  * Myeloid sarcoma, myeloid proliferations related to Down Syndrome, or blastic plasmacytoid dendritic cell neoplasm
  * AML with trilineage dysplasia
* AML with adverse cytogenetics (defined as -5/-5q; -7/-7q; abnormal 3q, 9q, 11q, 20q, 21q, or 17p; t[6;9]; t[9;22]; trisomy 8; trisomy 13, complex karyotypes [>= 3 unrelated abnormalities]),
* No hyperleukocytosis with >= 50,000 blasts/uL (leukapheresis or hydroxyurea allowed for cytoreduction immediately prior to the first dose of alvocidib)
* No active CNS leukemia
* ECOG performance status 0-2
* Serum creatinine =< 2.0 mg/dL
* ALT/AST =< 5 times upper limit of normal
* Bilirubin =< 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* No active uncontrolled infection
* Infection that is under active treatment allowed provided it is controlled with antibiotics
* No other life-threatening illness
* No mental deficits and/or psychiatric history that would preclude giving informed consent or following study requirements
* At least 24 hours since prior leukapheresis or hydroxyurea for cytoreduction
* Prior non-cytotoxic therapies (e.g., thalidomide or lenalidomide, interferon, cytokines, low-dose 5-azacytidine, or low-dose cytoxan) for MDS or MPD allowed
* Prior chemotherapy or bone marrow/stem cell transplantation for non-AML malignancy allowed
* No prior alvocidib
* No other concurrent chemotherapy, radiotherapy, or immunotherapy
* No other concurrent investigational or commercially-available antitumor therapies for AML
* LVEF >= 45%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Karp, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (2):
- United States (2):
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All newly diagnosed adults diagnosed with AML were considered for participation.Enrolled on study between November 20, 2008 and July 20, 2010.
Pre-assignment Details: 2 patients on each arm consented to study, but were screen failures and did not start treatment.
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 37 | 37
Completed | 37 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 30 | 57
  >=65 years | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (54) | 59 (53) | 60 (58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 33
  Male | 26 | 19 | 45
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Description: Bone marrow showing less than 5% leukemic blasts with normal maturation of all cell lines, an ANC of at least 1000/uL and a platelet count of 100,000/uL, absence of blast in peripheral blood, absence of identifiable leukemic cells in the bone marrow, clearance of disease-associated cytogenetic abnormalities, and clearance of any previously existing extramedullary disease. Repeat marrow confirmation 4-6 weeks following the marrow documenting CR is not required due to the need for continued treatment in CR.
Time Frame: 1 year
Population: 39 patients had been enrolled in each arm with two patients in each arm receiving incomplete therapy
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 37 | 37
participants | 24 | 29

2. Secondary Outcome: Number of Participants Experiencing Death From Any Cause Within 60 Days of Starting FLAM
Description: Toxicity defined as death from any cause within 60 days of starting FLAM.
Time Frame: 60 days
Population: 39 patients had been enrolled in each arm with two patients in each arm receiving incomplete therapy. Toxicity defined as death from any cause within 60 days of starting FLAM.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 37 | 37
Participants | 3 | 3

3. Secondary Outcome: Disease-free Survival
Description: This will be defined as the time between study entry and the first date that recurrent or progressive disease is objectively documented, or death from any cause occurs.
Time Frame: up to 2 years
Population: 39 patients had been enrolled in each arm with two patients in each arm receiving incomplete therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 37 | 37
months | 13.6 [10.1 to NA] — The 95% confidence interval is reported as 10.1 to infinity (10.1-inf) | 12.0 [9.2 to NA] — The 95% confidence interval is reported as 9.2 to infinity (9.2-inf)

ADVERSE EVENTS:
Time Frame: 1 cycle of therapy
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 8/39 | 8/39
Other Adverse Events (participants affected / at risk) | 1/39 | 1/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=39) | Arm II (N=39)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Oral and/or Gastrointestinal mucositis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Cardiac dysfunction (Cardiac disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=39) | Arm II (N=39)
General disorders-other (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less